CLINICAL TRIAL: NCT01947426
Title: Effect of Maternal Supplementation With DHA During Pregnancy and Lactation on the Development of the Term Newborn
Brief Title: Effect of Mother DHA Supplementation on Term Newborn.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Puleva Biotech (Industry)
Responsible Party: Principal Investigator, Julio J. Ochoa, Julio J. Ochoa, Professor, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C3565-00; C3565-00 (Other: Lactalis PULEVA)
Record Dates: First submitted 2013-09-04; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Oxidative Stress; Inflammation; Infant Development
Keywords: DHA, term neonates, mother milk
MeSH Terms: conditions — Inflammation | interventions — Docosahexaenoic Acids; Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA supplementation (Experimental): mother consuming 400 mg/day of DHA and tehir neonates
  Interventions: Dietary Supplement: DHA Supplementation
- Control (milk without DHA) (Placebo Comparator): Mothers comsuming placebo and their neonates
  Interventions: Dietary Supplement: Control (milk without DHA)

INTERVENTIONS:
Dietary Supplement: DHA Supplementation — mothers consuming 400 mg of DHA/day and their neonates
  Other Names: Docosahexaenoic acid
  Arms: DHA supplementation
Dietary Supplement: Control (milk without DHA) — mothers consuming placebo product and their neonates
  Other Names: Placebo group
  Arms: Control (milk without DHA)

SUMMARY:
In the present study, we evaluate the effect of the mother suplementación with DHA during the gestation and lactation on diverse aspects of the development of newborn. The effect on the oxidative stress, inflammatory signaling, bone turnover and piscomotor and visual development was studied. Women will in the sixth month of pregnancy, consume a diet balanced during last 3 months of pregnancy and the whole lactation. In addition the women will divide in two groups: one will receive a supplement of docosahexaenoic acid (DHA) to evaluate the effects on the development of the newborn child; whereas another group will receive a placebo. Different samples of blood of the mother and of mother milk will be taken and we will correlating her lipidic profile with the brain development of the newborn child, evaluated by different tests.

DETAILED DESCRIPTION:
The sample will be 120 volunteers that will be enrolled in the services of Gynaecology of the infantile Hospital of Granada. The pregnant women will be assigned from random form to one of 2 groups that are described later:

Group A: balanced diet Mediterranean, intake of 2 glasses / day of the dairy drink control.

Group B: balanced Mediterranean diet together with the consumption of 400mg/day of DHA in the dairy product (2 glasses / day). The dairy products will be distributed in white packages without any indication that reflects the type of product that contains (double blind). Every volunteer will be assigned a key that guarantees the confidentiality of their analytical values.

The dietary intervention will begin in the sixth month of pregnancy and will conclude to the third month of lactation (though there will improve itself the importance of a mother lactation up to 6 month postpartum). There will be obtained samples of blood (5 mL) of the mothers in the moment of the capture, in the childbirth and to 3 postpartum months. There will take a sample of blood of umbilical cord (5mL) in the moment of the childbirth (vein and artery). In addition there will take a sample of blood of the child (5mL) to 2.5 months. There will take also samples of mother milk (10mL), concretely of colostrum (2-3 postpartum days) and of mature(ripe) milk to 1, 2, 3 months. The samples will be preserved in freezer of-80ºC and sent to the different laboratories due preserved participants in order that there does not break the cold chain ( dry ice). In the first year of life of the child there will be practised tests of motive and cognitive development (Bayley's test and Fagan's test) in order to evaluate the influence of the dietetic intervention on the mother in the development of the child.

ELIGIBILITY:
Inclusion Criteria:

1. Consent
2. mother with normal gestation.

Exclusion Criteria:

1. Risk factors during gestation.
2. Lactose intolerance
3. systemic illness.
4. Kwashiorkor.
5. Metabolic illness.
6. Foetal pathologies

Max Age: 40 Years | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change of Visual Development of newborn | Change from Baseline at 12 months of life
  Visual Evoked Potentials

SECONDARY OUTCOMES:
Change of bone turnover biomarkers in blood samples during supplementation | Change from Baseline after supplementation (2,5 months)
  indicators of Bone turnover in the mother and their child
Change of oxidative stress parameters in mother milk samples during supplementation | Change from Baseline after supplementation (2,5 months)
  oxidative stress parameters (indicators of oxidative stress to lipids and proteins and antioxidant defense)
Motor and cognitive development of newborn | 12 months
  Bayleys test

CONTACTS AND LOCATIONS:
Overall Officials: Julio J Ochoa, Principal Investigator — Universidad de Granada
Locations (1):
- Julio J. Ochoa, Granada, Granada, Spain

REFERENCES:
- [Derived] Hurtado JA, Iznaola C, Pena M, Ruiz J, Pena-Quintana L, Kajarabille N, Rodriguez-Santana Y, Sanjurjo P, Aldamiz-Echevarria L, Ochoa J, Lara-Villoslada F; NUGELA Group. Effects of Maternal Omega-3 Supplementation on Fatty Acids and on Visual and Cognitive Development. J Pediatr Gastroenterol Nutr. 2015 Oct;61(4):472-80. doi: 10.1097/MPG.0000000000000864. PMID 25988553